CLINICAL TRIAL: NCT06963554
Title: Randomized Controlled Trial of Project Support
Brief Title: Examining Whether Project Support Works
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Caitlin Elizabeth Rancher, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00144297
Record Dates: First submitted 2025-04-25; First posted 2025-05-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-04

CONDITIONS: Parent-Child Relations; Parenting Self Efficacy; Child Mental Health
Keywords: Child trauma; Non-offending caregiver

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Support (Experimental): All participants will complete a baseline assessment on demographics, parenting behaviors, and mental health symptoms. Participants randomized to the experimental condition will receive Project Support and be offered case management services. Approximately 4-6 weeks after the baseline assessment all participants will complete a post-test assessment that includes measures of service satisfaction.
  Interventions: Behavioral: Project Support; Behavioral: Case Management Services
- Treatment as usual (Other): All participants will complete a baseline assessment on demographics, parenting behaviors, and mental health symptoms. Participants randomized to the treatment as usual condition will receive routine provision of case management services. Approximately 4-6 weeks after the baseline assessment all participants will complete a post-test assessment that includes measures of service satisfaction.
  Interventions: Behavioral: Case Management Services

INTERVENTIONS:
Behavioral: Project Support — The Project Support intervention involves up to four 60-minute individual counseling sessions focused on teaching caregivers how to listen to and comfort their child. Participants will receive didactic instruction and feedback on their use of the skills in role-plays with a treatment provider and with their child. In the role-plays the provider first demonstrates how to use the skill in a brief example of typical situations in which the skill could be used. In these examples the caregiver takes on the role of their child and the provider takes on the role of the caregiver. Subsequently the caregiver and provider switch roles so the caregiver has an opportunity to practice executing the skill. The provider helps the caregiver process their experience of each role-play and provides real-time, targeted feedback to help the caregiver develop their ability to use the skills.
  Arms: Project Support
Behavioral: Case Management Services — Case management services, or treatment as usual, may involve referrals for financial resources or donated goods, as well as assistance with court, law enforcement, or information about orders of protection. The nature of these services depends on the needs identified by the family and case manager. There is currently no standard "treatment" offered to families on the waitlist. This condition will receive individually tailored services, as needed.

SUMMARY:
This study will involve a randomized, controlled trial with two parallel groups, Project Support and a treatment as usual control group. Families with a child on the waitlist for trauma-focused services will be invited to participate. Participation involves completing a baseline assessment of family functioning and trauma characteristics. Participants will then be randomized to either Project Support or the treatment as usual control group. All participants will be invited to complete the post-test assessment 4-6 weeks after the baseline assessment, prior to beginning trauma-focused services.

DETAILED DESCRIPTION:
The proposed research addresses the dearth of brief, empirically-supported programs designed for caregivers to mitigate the adverse effects of child trauma. This project will examine the telehealth delivery of Project Support, a program that addresses parenting skills and behavior problems among children exposed to violence or maltreatment. Project Support uses didactic, tailored instruction to teach caregivers how to listen to and comfort their child. This study builds on prior research which has found that Project Support is feasible and acceptable for both treatment providers and families on the waitlist for trauma-focused services. This phase of the research will examine the preliminary efficacy of Project Support in a randomized controlled trial, evaluating the impact of this intervention on caregiver emotional support, parenting self-efficacy, and family distress, compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Family is seeking trauma-focused services for their child;
* Child is between 6 - 13 years old;
* Caregiver agreed to be contacted for volunteer research opportunities;
* Caregiver and child can communicate in English;
* Child has been living with caregiver for at the last 6 months or longer;
* Family is able to participate in services delivered via telehealth.

Exclusion Criteria:

* Child or caregiver has a diagnosis that would impair their ability to participate in or benefit from services (e.g., traumatic brain injury, developmental disability, psychosis);
* Child is in Foster Care or Department of Social Services custody;
* The caregiver is unwilling or unable to give informed consent and/or the child is unwilling and unable to give assent.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Parenting self-efficacy assessed by the Tool to Measure Parenting Self-Efficacy (TOPSE) | Baseline to Post-test (6 weeks)
  Caregivers will complete the Tool to Measure Parenting Self-Efficacy (TOPSE). Responses to this questionnaire assess several domains of parenting. Responses to items assessing parenting self-efficacy (e.g., "I am able to comfort my child") are made on a 11-point scale (0 = completely disagree, 10 = completely agree). Responses are summed to create a total score. This outcome measure will be assessed by comparing both within- and between-person changes in parenting self-efficacy from baseline to post-test.
Supportive parenting assessed by the Parent Behavior Inventory | Baseline to Post-test (6 weeks)
  Caregivers and children will complete convergent versions of the Parent Behavior Inventory. Responses to this questionnaire assess several domains of parenting. Responses to items assessing supportive/engaged parenting (e.g., "I listen to ___'s feelings and try to understand them") are made on a 6-point scale (0 = not at all true to 5 = very true). Responses are summed to create a total score. This outcome measure will be assessed by comparing within- and between-person changes in supportive parenting from baseline to post-test.
Attendance to trauma-focused treatment intake session coded from clinical records | 4 months after Post-test
  Research staff will review clinical records to determine whether participants attended their intake session. This will be coded dichotomously as whether or not the family attends the intake appointment ( 0 = did not attend intake, 1 = attended intake). Families will be determined to have attended their intake if this is noted either in clinic records as "in treatment" or if there is an "intake note" available in the clinical record. We will monitor the status of intake attendance for up to 4 months after the family completes participation in the post-test assessment.

SECONDARY OUTCOMES:
Child psychological distress assessed by the Pediatric Symptom Checklist | Baseline to Post-test (6 weeks)
  Caregivers and children will complete convergent versions of the Pediatric Symptom Checklist. Responses to items on this questionnaire measuring child psychological distress (e.g., "Feels sad, unhappy") are made on a 3-point scale (0 = never, 1 = sometimes, 2 = often). Responses are summed to create a total score, with higher scores indicating greater psychological distress. This outcome measure will be assessed by comparing within and between-person changes in child psychological distress from baseline to post-test.
Child self-blame appraisals assessed by the Child Attributions and Perceptions Scale (CAPS) | Baseline to Post-test (6 weeks)
  Children will complete the Child Attributions and Perceptions Scale (CAPS) assessing their self-blame appraisals (e.g., "Do you blame yourself when things go wrong?") on a 5-point scale (1 = never to 5 = always). Responses are summed to create a total score, with higher scores indicating greater self-blame. This outcome measure will be assessed by comparing within- and between-person change from baseline to post-test.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Rancher, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No